CLINICAL TRIAL: NCT02637427
Title: Does Plasma Reduce Bleeding in Patients Undergoing Invasive Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Pittsburgh (Other); Johns Hopkins University (Other); University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro20150001801; 1R34HL125804-01A1 (NIH)
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Blood Coagulation Disorders; Hemorrhage
Keywords: Fresh frozen plasma; Bleeding
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fresh frozen plasma transfusion (Experimental): Pre-procedure fresh frozen plasma transfusion (15 cc per Kg, range 10-20 cc/Kg, to a maximum of 5 units)
  Interventions: Biological: Fresh frozen plasma transfusion
- No transfusion (No Intervention): No transfusions prior to the procedure

INTERVENTIONS:
Biological: Fresh frozen plasma transfusion — Pre-procedure fresh frozen plasma transfusion (15 cc per Kg to a maximum of 5 units)
  Arms: Fresh frozen plasma transfusion

SUMMARY:
The purpose of this study is to evaluate prophylactic fresh frozen plasma transfusion in patients with moderately elevated international normalized ratios (INR) prior to undergoing an invasive procedure.

DETAILED DESCRIPTION:
Fresh frozen plasma is used very frequently in the US. Many plasma transfusions are given prior to a procedure in order to correct perceived bleeding risk, yet there is little evidence to support that use of plasma reduces bleeding. There has never been an adequately powered trial to establish the efficacy of plasma and document the risks. This pilot study will evaluate the feasibility of conducting a research protocol that will lead to a large scale clinical trial designed to evaluate the treatment effectiveness of prophylactic plasma transfusion in patients with moderately elevated INRs prior to undergoing an invasive procedure outside of the operating room.

Study subjects will be randomly allocated to either receive either plasma transfusion prior to the procedure, or to no treatment. Study outcomes will be compared between the two study arms. Recruitment rates, protocol adherence, and rates of study outcomes will be assessed to determine the feasibility of the large scale trial.

ELIGIBILITY:
Inclusion Criteria:

1. INR level between 1.50 and 2.50 inclusive
2. undergoing an invasive procedure at the bedside, endoscopy laboratory, or in radiology

Exclusion Criteria:

1. undergoing a surgical procedure in the operating room;
2. active bleeding;
3. undergoing a procedure involving or proximal to the central nervous system or spinal cord;
4. cardiac catheterization,
5. using 4 factor plasma concentrates
6. using systemic heparin/heparinoid therapy, direct factor X inhibitors and other anticoagulants for which plasma will not correct prolonged INR;
7. platelet count less than 50,000/ul,
8. congenital coagulation disorders;
9. acquired disorders (i.e., lupus anticoagulant) for which plasma will not correct the disorder;
10. women who are pregnant and;
11. unwillingness to consider blood transfusion.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Study Chair — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - Johns Hopkins University, The Johns Hopkins Hospital, Baltimore, Maryland
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Started | 27 | 30
Completed | 27 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (18.0) | 58.2 (13.9) | 56.0 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 16 | 21 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 57
Liver disease [Count of Participants; unit: Participants] | 15 | 22 | 37
Hypertension [Count of Participants; unit: Participants] | 14 | 19 | 33
Diabetes [Count of Participants; unit: Participants] | 10 | 14 | 24
Coronary artery disease [Count of Participants; unit: Participants] | 4 | 7 | 11
Congestive heart failure [Count of Participants; unit: Participants] | 3 | 9 | 12
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants] | 1 | 3 | 4
Thromboembolism [Count of Participants; unit: Participants] | 4 | 1 | 5
Prior history of bleeding [Count of Participants; unit: Participants] | 6 | 2 | 8
Metastatic carcinoma [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin Level
Description: Change from pre-procedure hemoglobin to lowest within 2 days after procedure
Time Frame: within 2 days post procedure
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
g/dL | -0.6 (1.0) | -0.4 (0.6)

2. Secondary Outcome: Number of Red Blood Cell Transfusions
Description: Differences in number of units of red blood cell transfusions between the two study arms
Time Frame: within 2 days post procedure
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
units | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Number of Participants With Transfusion Associated Cardiac Overload (TACO)
Description: Difference in rates between the two study arms
Time Frame: within 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
Participants | 0 | 2

4. Secondary Outcome: Number of Participants With Transfusion Related Acute Lung Injury (TRALI).
Description: Difference in rates between the two study arms
Time Frame: with 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Major Bleed
Description: 2g/dL or greater fall in hemoglobin level
Time Frame: with 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
Participants | 1 | 0

6. Secondary Outcome: Change in International Normalized Ratio (INR) Level Post Procedure
Description: Change from pre-procedure INR level
Time Frame: day of procedure
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 19 | 20
ratio | -0.24 (0.26) | 0 (0.15)

7. Secondary Outcome: Change in INR Level Day 1
Description: Change from pre-procedure INR level
Time Frame: day 1 post procedure
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 25 | 27
ratio | -0.22 (0.19) | -0.03 (0.19)

8. Secondary Outcome: Change in INR Level Day 2
Description: Change from pre-procedure INR level
Time Frame: day 2 post procedure
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 22 | 20
ratio | -0.09 (0.39) | 0 (0.19)

9. Secondary Outcome: Mortality (Number of Participants)
Description: Death
Time Frame: in-hospital up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With Infection
Description: Pneumonia or blood stream infection
Time Frame: within 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
Participants
  Pneumonia | 0 | 1
  Blood stream infection | 2 | 1

11. Secondary Outcome: Number of Participants With ICU Admission
Description: new admission to the intensive care unit
Time Frame: within 2 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
Number analyzed (Participants) | 27 | 30
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: In-hospital (for up to 7 days)
Description: Adverse events were captured via daily medical record review
Arm/Group | Fresh Frozen Plasma Transfusion | No Transfusion
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/27 | 3/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fresh Frozen Plasma Transfusion (N=27) | No Transfusion (N=30)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2)
Blood Stream Infrection (Infections and infestations) | 2 (2) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT02637427/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT02637427/ICF_001.pdf